CLINICAL TRIAL: NCT07100860
Title: Does Duration Matter? A Study on Single-Lung Ventilation Time and Pulmonary Complications in Thoracic Procedures
Brief Title: The Effect of Single Lung Ventilation Duration on Postoperative Pulmonary Complications in Thoracic Surgery
Status: Recruiting | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ekin Guran, MD, Consultant Anesthesiologist, Ankara Etlik City Hospital
Other Study IDs: OLV_PPC
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pulmonary Complications; One Lung Ventilation; Ards; Postoperative Pulmonary Atelectasis
Keywords: postoperative pulmonary complications; one lung ventilation
MeSH Terms: conditions — Acute Lung Injury; Pulmonary Atelectasis | interventions — One-Lung Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: One-Lung ventilation — In this observational study, the naturally occurring duration of intraoperative single-lung ventilation (SLV) during thoracic surgery will be recorded. No intervention is applied or modified for research purposes. The exposure of interest is the total duration (in minutes) of SLV, which will be timed from initiation to termination during surgery. This variable will be analyzed in relation to postoperative pulmonary complications.

SUMMARY:
This observational study investigates the relationship between the duration of single-lung ventilation (SLV) and the incidence of postoperative pulmonary complications (PPCs) such as pneumonia, pneumothorax, hemothorax, acute lung injury, and acute respiratory distress syndrome (ARDS) in adult patients undergoing thoracic surgery. A total of 134 patients aged 18-85 years, scheduled for thoracic surgery requiring SLV, will be monitored. Data including SLV duration, perioperative parameters, and postoperative pulmonary outcomes will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years Undergoing thoracic surgery OLV planned during the procedure

Exclusion Criteria:

Pediatric patients Patients not requiring OLV Previous thoracic surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 to 85 years who are scheduled to undergo thoracic surgery at Etlik City Hospital and require OLV during the procedure. Patients will be included if they meet the eligibility criteria of being over 18 years old, undergoing thoracic surgery, receiving intraoperative OLV, and providing informed consent to participate in the study. Patients will be excluded if they are part of the pediatric age group, do not require OLV, or decline participation. A total of 134 eligible patients will be prospectively enrolled and followed for seven days postoperatively to assess the occurrence of pulmonary complications.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Postopertive Pulmonary Complications | postoperative 7 days
  Postoperative pulmonary complications (PPCs) are defined as respiratory events occurring within the first seven days following thoracic surgery, which negatively impact patient outcomes. In this study, PPCs include pneumonia, pneumothorax, hemothorax, acute lung injury, acute respiratory distress syndrome (ARDS), prolonged oxygen requirement, unplanned reintubation, and the need for non-invasive ventilation. These complications will be identified through clinical assessment, arterial blood gas analysis, and postoperative imaging such as chest X-rays. Each case will be evaluated using predefined diagnostic criteria to ensure consistency. The incidence of PPCs will be analyzed in relation to the duration of intraoperative single-lung ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Hazal EG AYTUĞ, Study Director — Consultant Anesthesiologist
Locations (1):
- Hazal Ekin GÜRAN AYTUĞ, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Kiss T, Bluth T, Gama de Abreu M. [Does intraoperative lung-protective ventilation reduce postoperative pulmonary complications?]. Anaesthesist. 2016 Aug;65(8):573-9. doi: 10.1007/s00101-016-0198-8. German. PMID 27392439